CLINICAL TRIAL: NCT06115447
Title: Polypropylene vs Polyglactin in Suturing of the Lung
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Younus, Principle investigator, Assiut University
Other Study IDs: polyglactin lung suturing
Record Dates: First submitted 2023-10-11; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Lung Injury; Bleb Lung; Lung Cancer
MeSH Terms: conditions — Lung Injury; Blister; Lung Neoplasms | interventions — Polyglactin 910; Polypropylenes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polyglactin group: lung suturing with polyglactin
  Interventions: Procedure: lung suturing with polyglactin
- Polypropylene Arm: lung suturing with Polypropylene
  Interventions: Procedure: ung suturing with polypropylene

INTERVENTIONS:
Procedure: lung suturing with polyglactin — lung suturing with polyglactin
  Groups: Polyglactin group
Procedure: ung suturing with polypropylene — ung suturing with polypropylene
  Groups: Polypropylene Arm

SUMMARY:
Comparative study comparing polypropylene and Polyglactin in suturing of the lung

DETAILED DESCRIPTION:
Lung tear or, pulmonary laceration is an injury in lung parenchyma, said injury can be caused by several reasons:

Blunt chest trauma Penetrating trauma such as stab wounds or firearm wounds Iatrogenic, such as faulty intercostal tube insertion

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Assiut University Hospital And will undergo surgery for lung tear repair.
* Patients admitted to Assiut University Hospital And will undergo surgery for bullectomy or lobectomy.

Exclusion Criteria:

* Patients with lung injury repaired with a stapler

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presented to cardiothoracic surgery department and trauma department with the inclusion criteria applied
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
duration in days of intercostal tube air leak with each group | 2 weeks
  Polypropylene vs Polyglactin

REFERENCES:
- [Background] Regan T, Lawrence N. Comparison of poliglecaprone-25 and polyglactin-910 in cutaneous surgery. Dermatol Surg. 2013 Sep;39(9):1340-4. doi: 10.1111/dsu.12265. Epub 2013 Aug 13. PMID 23941601
- [Background] Rendeki S, Molnar TF. Pulmonary contusion. J Thorac Dis. 2019 Feb;11(Suppl 2):S141-S151. doi: 10.21037/jtd.2018.11.53. PMID 30906578
- [Background] Romby P, Carbon P, Westhof E, Ehresmann C, Ebel JP, Ehresmann B, Giege R. Importance of conserved residues for the conformation of the T-loop in tRNAs. J Biomol Struct Dyn. 1987 Dec;5(3):669-87. doi: 10.1080/07391102.1987.10506419. PMID 3078237